CLINICAL TRIAL: NCT05977192
Title: Mobile Health-based Motivational Interviewing to Promote Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Vaccination in Oklahomans
Brief Title: Mobile Health-based Motivational Interviewing to Promote COVID-19 Vaccination
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Ashlea Braun, Assistant Professor, Oklahoma State University Center for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-282-STW
Record Dates: First submitted 2023-07-30; First posted 2023-08-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard MI (Experimental)
  Interventions: Behavioral: Standard MI; Behavioral: Ecological momentary assessment (EMA) messages
- Intensive MI (Experimental)
  Interventions: Behavioral: Intensive MI; Behavioral: Ecological momentary assessment (EMA) messages
- MOTIVACC (Experimental)
  Interventions: Behavioral: MOTIVACC; Behavioral: Ecological momentary assessment (EMA) messages

INTERVENTIONS:
Behavioral: Standard MI — One phone-based MI session
  Arms: Standard MI
Behavioral: Intensive MI — Four phone-based MI sessions
  Arms: Intensive MI
Behavioral: MOTIVACC — mHealth-based MI
  Arms: MOTIVACC
Behavioral: Ecological momentary assessment (EMA) messages — EMA messages focused on vaccinations and health

SUMMARY:
The objective of this study is to evaluate the preliminary efficacy and acceptability of an mobile Health-based motivational interviewing (MI) intervention to promote SARS-CoV-2 vaccination (MOTIVACC) compared to traditional phone-based MI.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Reside in a rural area
* No previous dose of a SARS-CoV-2 vaccine
* Speak English
* Able to provide informed consent

Exclusion Criteria:

* A cognitive or other disability that inhibits smart phone use
* Inability to participate because of medical or psychiatric conditions diagnosed by a physician/clinician
* Enrollment in other COVID-19 research; pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in vaccine hesitancy and confidence | Baseline and follow-up (8 weeks)
Changes in intention to receive the vaccine | Baseline and follow-up (8 weeks)

SECONDARY OUTCOMES:
Changes in expectations related to vaccines | Baseline and follow-up (8 weeks)
Changes in self-efficacy | Baseline and follow-up (8 weeks)
Changes in ambivalence | Baseline and follow-up (8 weeks)
Changes in value-behavior discrepancy | Baseline and follow-up (8 weeks)
Number of participants who receive the COVID-19 vaccine | Follow-up (8 weeks)

OTHER OUTCOMES:
Percentage of total of ecological momentary assessment messages opened/viewed | 8 weeks (from baseline to follow up)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma State University, Stillwater, Oklahoma

REFERENCES:
- [Derived] Braun A, Corcoran S, Tu Doan K, Jernigan C, Moriasi C, Businelle M, Bui T. Mobile Health-Based Motivational Interviewing to Promote SARS-CoV-2 Vaccination in Rural Adults: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 28;14:e64010. doi: 10.2196/64010. PMID 40294409